CLINICAL TRIAL: NCT06427122
Title: The Effect of the EMD Protocol for Urge Compared to Care as Usual on Dermatology-specific Quality of Life
Brief Title: Effect of EMD Protocol for Urge on Dermatology-specific Quality of Life
Acronym: EMD-U vs CAU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tamar Nijsten (Other)
Responsible Party: Sponsor-Investigator, Tamar Nijsten, Prof., Erasmus Medical Center
Organization: Erasmus Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11074; NL84417.078.23 (Other: ToetsingOnline)
Record Dates: First submitted 2024-02-07; First posted 2024-05-23 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Atopic Dermatitis; Prurigo Nodularis
Keywords: EMD Protocol for Urge; Quality of Life; Itch; Scratching
MeSH Terms: conditions — Dermatitis, Atopic; Pruritus

STUDY DESIGN:
Intervention Model Description: An open randomised controlled trial, with two arms: 1) EMD-U, 2) CAU (control).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMD-U (Experimental): The EMD-U treatment lasts eight weeks, in which two EMD-U sessions of 60 minutes and two phone calls take place in the first three weeks. In the five following weeks, patients are phoned twice to ask for their experiences with the practicing at home. An important part of EMD-U consists of homework exercises. These homework exercises comprise to practice/apply the intervention as learned during the sessions with the therapist, in those situations wherein the urge to scratch their skin is present. In the text below, we will explain in more detail what the treatment protocol entails. Patients in this condition receive the EMD-U treatment in addition to the care as usual.
  Interventions: Behavioral: EMD Protocol for Urge; Other: Care as Usual
- Care as Usual (Active Comparator): Patients in the control group receive care as usual (CAU), which is the standard care of the dermatologist. In addition to completing the questionnaires at T0, 1, 2, 3, and 4 these patients are not offered any additional treatment or support aimed at their scratching behaviour.
  Interventions: Other: Care as Usual

INTERVENTIONS:
Behavioral: EMD Protocol for Urge — During the EMD-U sessions, the patient is asked to focus on the spot on his/her skin where the urge to scratch is highest. The patient is asked to rate the level of urge to scratch this spot on a 10-point scale and to imagine that they scratch this spot as they would like. At the same time eye movements are offered for 30 seconds. This procedure is repeated until the level of urge to scratch has become nihil. This procedure is repeated for all other skin parts where the patient experiences an urge to scratch, until there are no skin parts left. As a homework assignment straight after the first session, the patient is instructed and encouraged to practice the same intervention at home. The two EMD-U sessions and two phone calls, take place in the first three weeks of the study. In the five following weeks, patients are phoned twice to ask for their experiences with the practicing at home.
  Arms: EMD-U
Other: Care as Usual — Patients in the control group receive care as usual (CAU), which is the standard care of the dermatologist. In addition to completing the questionnaires at T0, 1, 2, 3, and 4 these patients are not offered any additional treatment or support aimed at their scratching behaviour.

SUMMARY:
The primary objective of this open randomised controlled trial is to assess the add-on effect of EMD-U compared to CAU alone, in improving dermatology-specific quality of life in patients with atopic dermatitis or prurigo nodularis who suffer from severe scratching behaviour.

The main study parameter is the difference in treatment effect between EMD-U and CAU at T2, measured with the Skindex-29 symptoms scale. There are five measurement points: T0, T1 after 4 weeks, T2 after 8 weeks, T3 after 12 weeks, and T4 after 6 months.

Patients are randomly allocated to either the EMD-U or CAU condition.

DETAILED DESCRIPTION:
Rationale: The EMD protocol for urge (EMD-U) is a recently developed treatment that combines elements of Eye Movement Desensitization and Reprocessing (EMDR) therapy, Cognitive Behaviour therapy, and hypnotherapy. EMD-U aims to reduce the urge for scratching behaviour through desensitization techniques, self-registration of behaviour, and homework assignments. The EMD-U treatment has shown promising results in reducing scratching behaviour in patients with atopic dermatitis and is currently being investigated in patients with prurigo nodularis. Yet, the added value of the brief EMD-U intervention in addition to the care as usual (CAU) in improving dermatology-specific quality of life is unknown.

Objective: The primary objective of the study is to assess the add-on effect of EMD-U compared to CAU alone, in improving dermatology-specific quality of life in patients with atopic dermatitis or prurigo nodularis who suffer from severe scratching behaviour.

Study design: An open randomised controlled trial, with two arms: 1) EMD-U, 2) CAU (control). There are five measurement points: T0, T1 after 4 weeks, T2 after 8 weeks, T3 after 12 weeks, and T4 after 6 months.

Study population: Patients with atopic dermatitis or prurigo nodularis who suffer from substantial scratching behaviour.

Intervention (if applicable): Patients are randomly allocated to either the EMD-U or CAU condition.

The EMD-U treatment lasts eight weeks, in which two EMD-U sessions and two phone calls take place in the first three weeks. After the first EMD-U session, patients are instructed to apply the learned technique at home until the end of the study. In the five following weeks, patients are phoned twice to ask for their experiences with the practicing at home.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 ≥
* A confirmed diagnosis of atopic dermatitis or prurigo nodularis
* Suffering from persistent and frequent scratching behaviour
* IGA-CPG activity score ≥ 3 OR Skindex-29 symptoms subscale score ≥ 42
* Stable course of treatment in the two weeks prior to the study (no medication change, etc.)
* Sufficiently motivated to take part in a new intervention aimed at behaviour change

Exclusion Criteria:

* Insufficient understanding of Dutch language
* Severe psychiatric disorders that require treatment first, such as delusional disorder or major depression
* If medication is changed during the course of the study, the participant will be considered a drop-out from the moment the medication has changed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2024-03-11 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Skindex-29 | measured at the start of the study (T0), in week 4 (T1), in week 8 (T2), and during follow-up, in week 12 (T3) and six months after T0 (T4).
  The main study outcome is the dermatology-specific health-related quality of life (HRQOL). It consists of 30 items to be scored on a 5-point response scale. Outcome ranges from 0 (never) to 100 (all the time). The sum of scores is devided by the number of items answered. Higher scores indicate worse quality of life. The instrument has three subscales: symptoms, emotions, and functioning.

SECONDARY OUTCOMES:
Eczema Area and Severity Index (EASI) | Measured at the start of the study (T0), in week 4 (T1), in week 8 (T2), and during follow-up, in week 12 (T3) and six months after T0 (T4).
  This is a validated scoring system that grades the physical signs of atopic dermatitis/eczema.
  The minimum EASI score is 0 and the maximum EASI score is 72. Higher scores indicate higher disease activity.
Investigator Global Assessment (IGA) | Measured at the start of the study (T0), in week 4 (T1), in week 8 (T2), and during follow-up, in week 12 (T3) and six months after T0 (T4).
  The IGA is a 5-point tool for the objective assessment of chronic prurigo. The IGA for stage of chronic nodular prurigo (CNPG) and signs of activity in chronic prurigo are used. Items range from 0 (clear) to 4 (severe). Higher scores indicate higher disease activity.
EQ-5D-5L | Measured at the start of the study (T0), in week 4 (T1), in week 8 (T2), and during follow-up, in week 12 (T3) and six months after T0 (T4).
  It is a generic instrument that can be used in a wide range of health conditions and treatments. The EQ-5D-5L consists of a descriptive system and the EQ VAS. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale.
  Health state index scores generally range from less than 0 (where 0 is the value of a health state equivalent to dead; negative values representing values as worse than dead) to 1 (the value of full health), with higher scores indicating higher health utility. The visual analogue scale (VAS), on which the patient rates his/her perceived health, ranges from 0 (the worst imaginable health) to 100 (the best imaginable health).
The Self-Control Cognition Questionnaire, Dutch: Zelfcontrole Cognitie Vragenlijst (ZCCL) | Measured at the start of the study (T0), in week 4 (T1), in week 8 (T2), and during follow-up, in week 12 (T3) and six months after T0 (T4).
  The ZCCL is an 11-item self-report questionnaire measuring perceived self-control. There are two subscales: 'positive reward' (of the unwanted behaviour) and 'difficulty resisting'. Each item is scored on a 5-point Likert scale, ranging from 1 (not applicable at all) to 5 (totally applicable). Total score ranges from 11-55. Higher scores indicate less self-control.
Patient Health Questionnaire for anxiety and depression (PHQ-4) | Measured at the start of the study (T0), in week 4 (T1), in week 8 (T2), and during follow-up, in week 12 (T3) and six months after T0 (T4).
  The PHQ-4 is a brief self-report screening tool for depression and anxiety, consisting of four items. Two items on depression, and two items on anxiety are scored with a 4-point Likert scale, ranging from 0 (not at all) to 3 (nearly every day). Higher scores indicate more depression and anxiety symptoms.
Skin Picking Scale (SPS) | Measured at the start of the study (T0), in week 4 (T1), in week 8 (T2), and during follow-up, in week 12 (T3) and six months after T0 (T4).
  a six-item self-report measure for the assessment of skin picking behaviour. The scale has a total score range of 0-24. Higher scores indicate more skin picking.

OTHER OUTCOMES:
Life Events Checklist for DSM-5 (LEC-5) | At start of study (T0)
  The LEC-5 is a 17-item self-report questionnaire designed to screen for potentially traumatic events in a respondent's lifetime. It identifies whether the person has gone through any of the listed events, and there is no definitive scoring procedure or interpretation involved. Respondents indicate varying levels of exposure to each type of potentially traumatic event included on a 6-point nominal scale, and respondents may endorse multiple levels of exposure to the same trauma type. The LEC-5 does not yield a total score or composite score.
Treatment Expectation Questionnaire (TEX-Q) | At start of study (T0)
  The TEX-Q is a 15-item self-report questionnaire assessing patients' expectations of medical and psychological treatments. The scale of the items ranges from 0 to 10. Higher scores indicate higher expectations. The English version of the TEX-Q will be translated into Dutch, using the FACIT translation methodology.
Mental imagery | At start of study (T0)
  patients are requested to assess their capacity for engaging in visuomotor activities through mental imagery, utilizing a 4-point Likert scale ranging from 0 (totally disagree) to 3 (totally agree). A higher score indicates better imagination capacity.
Visits | Six months after start study (T4)
  Number of hospital visits and medication

CONTACTS AND LOCATIONS:
Overall Officials: Rick Waalboer-Spuij, MD, PhD, Principal Investigator — Erasmus University Medical Center, Department of Dermatology; Leonieke W Kranenburg, PhD, Principal Investigator — Erasmus University Medical Center, Department of Psychiatry, Section Medical Psychology
Locations (1):
- Erasmus University Medical Center, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No
No IPD is shared due to privacy issues

REFERENCES:
- [Background] de Veer MR, Waalboer-Spuij R, Hijnen DJ, Doeksen D, Busschbach JJ, Kranenburg LW. Reducing scratching behavior in atopic dermatitis patients using the EMDR treatment protocol for urge: A pilot study. Front Med (Lausanne). 2023 Apr 4;10:1101935. doi: 10.3389/fmed.2023.1101935. eCollection 2023. PMID 37081840